## Study method and statistical analysis

The couples included in the study were divided into two groups: study and control groups. All patients completed the demographic information scale, The COMPI Coping Strategy Scales, Golombok Rust Sexual Satisfaction Scale and Marital Adjustment Scale. Back massage was taught to the couples in the study group and the spouses were allowed to perform back massage during the infertility treatment. No intervention was applied in the control group. A month later, the COMPI Coping Strategy Scales, Golombok Rust Sexual Satisfaction Scale and Marital Adjustment Scale were repeated on the fences.

The data were analyzed in the SPSS program. Catagorical variables were compared with the chi-square test and Fisher's extract test. For the analysis of continuous variables, t-test and Mann-Whitney u test were applied to independent variables. Wilcoxon test was applied in the analysis of dependent variables. p<0.005 was accepted as the significance level.

